CLINICAL TRIAL: NCT05078827
Title: A Randomized, Double-blind, Multi-center, Three-arm, Parallel-group, Multiple-dose, Placebo Controlled Study to Assess the Therapeutic Equivalence of Fluorouracil Cream USP 5% of Encube Ethicals Pvt. Ltd., India Compared With Fluorouracil 5% Topical Cream of Mylan Pharmaceuticals Inc., Morgantown, WV 26505 U.S.A. in the Treatment of Actinic Keratosis
Brief Title: Therapeutic Equivalence of Fluorouracil Cream, 5% Compared With Fluorouracil 5% Topical Cream of MylanPharmaceuticals Inc., U.S.A in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encube Ethicals Pvt. Ltd. (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBCC/2021/012
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Comparator Arm (Active Comparator): Reference Product (B): Fluorouracil 5% Topical Cream of Mylan Pharmaceuticals Inc., Morgantown, WV 26505 U.S.A.
  Interventions: Drug: Reference Product (B): Fluorouracil 5% Topical Cream of Mylan Pharmaceuticals Inc., Morgantown, WV 26505 U.S.A.
- Arms and Interventions (Experimental): Test Product (A): Fluorouracil Cream, 5% of Encube Ethicals Pvt. Ltd., India
  Interventions: Drug: Test Product (A): Fluorouracil Cream, 5% topical cream
- Placebo Arm (Placebo Comparator): Placebo Product (C): Test vehicle cream for fluorouracil 5% of Encube Ethicals Pvt. Ltd., India
  Interventions: Drug: Placebo Product (C): Test vehicle cream for fluorouracil 5% of Encube Ethicals Pvt. Ltd., India

INTERVENTIONS:
Drug: Test Product (A): Fluorouracil Cream, 5% topical cream — Apply cream twice daily in an amount sufficient to cover the lesions. Fluorouracil should be applied preferably with a nonmetal applicator or suitable glove. If Fluorouracil is applied with the fingers, the hands should be washed immediately afterward.
  Other Names: Experimental
  Arms: Arms and Interventions
Drug: Reference Product (B): Fluorouracil 5% Topical Cream of Mylan Pharmaceuticals Inc., Morgantown, WV 26505 U.S.A. — Apply cream twice daily in an amount sufficient to cover the lesions. Fluorouracil should be applied preferably with a nonmetal applicator or suitable glove. If Fluorouracil is applied with the fingers, the hands should be washed immediately afterward.
  Other Names: Active Comparator
  Arms: Comparator Arm
Drug: Placebo Product (C): Test vehicle cream for fluorouracil 5% of Encube Ethicals Pvt. Ltd., India — Apply cream twice daily in an amount sufficient to cover the lesions. Fluorouracil should be applied preferably with a nonmetal applicator or suitable glove. If Fluorouracil is applied with the fingers, the hands should be washed immediately afterward.
  Other Names: Placebo Comparator
  Arms: Placebo Arm

SUMMARY:
Fluorouracil is recommended for the topical treatment of multiple actinic or solar keratoses. In the 5% strength, it is also useful in the treatment of superficial basal cell carcinomas when conventional methods are impractical, such as with multiple lesions or difficult treatment sites.

DETAILED DESCRIPTION:
There is evidence that the metabolism of Fluorouracil in the anabolic pathway blocks the methylation reaction of deoxyuridylic acid to thymidylic acid. In this manner, Fluorouracil interferes with the synthesis of deoxyribonucleic acid (DNA) and to a lesser extent inhibits the formation of ribonucleic acid (RNA). As DNA and RNA are essential for cell division and growth, the effect of Fluorouracil may be to create a thymine deficiency, which, provokes unbalanced growth and death of the cell. The effects of DNA and RNA deprivation are most marked on those cells that grow more rapidly and take up Fluorouracil at a more rapid rate. The catabolic metabolism of Fluorouracil results in degradation products (e.g., CO2, urea, α-fluoro-β-alanine), which are inactive.

Systemic absorption studies of topically applied Fluorouracil have been performed on patients with actinic keratoses using tracer amounts of 14C-labeled Fluorouracil added to a 5% preparation. All patients had been receiving nonlabeled Fluorouracil until the peak of the inflammatory reaction occurred (2 to 3 weeks), ensuring that the time of maximum absorption was used for measurement. One gram of labeled preparation was applied to the entire face and neck and left in place for 12 hours. Urine samples were collected. At the end of 3 days, the total recovery ranged between 0.48% and 0.94%, with an average of 0.76%, indicating that approximately 5.98% of the topical dose was absorbed systemically. If applied twice daily, this would indicate systemic absorption of topical Fluorouracil to be in the range of 5 to 6 mg per daily dose of 100 mg. In an additional study, negligible amounts of labeled material were found in plasma, urine, and expired CO2 after 3 days of treatment with topically applied 14C-labeled Fluorouracil.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide voluntary informed consent and follow the protocol requirements
* Males or females at least 18 years of age
* Subjects with at least five (5) and no more than ten (10) clinically typical, visible, discrete, AK lesions, each at least 4 mm in diameter on the face or bald scalp. In this interpretation, if the total number of lesions on the face and bald scalp exceeds 10 and there are either 5-10 lesions on the face or 5-10 lesions on the bald scalp then select the designated treatment area that has 5-10 lesions (i.e., face or bald scalp)
* Skin pigmentation (Fitzpatrick skin type I, II, and III) that will allow differentiation of erythema assessment
* Females of childbearing potential must not be pregnant or lactating at Visit 1 (as confirmed by a negative urine pregnancy test with a sensitivity of less than 50 mIU/mL or equivalent units of human chorionic gonadotropin)
* Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, intrauterine device, a double barrier method, oral, transdermal, injected, or implanted nonhormonal or hormonal contraceptive) throughout the study. Female patients using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days before Visit 1 and should not change this regimen during the study. A sterile sexual partner is not considered an adequate form of birth control.

Exclusion Criteria:

* Known hypersensitivity or allergy to Fluorouracil or any of the excipients in the Test, Reference or Placebo products
* Presence of atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, or other possible confounding skin conditions on the face or bald scalp
* Use within 6 months before Visit 1 on the face or bald scalp of 1) chemical peel, 2) dermabrasion, 3) laser abrasion, 4) PUVA (psoralen plus ultraviolet A) therapy, or 5) ultraviolet B therapy
* Use within 1 month before Visit 1 on the face or scalp of 1) cryo destruction or chemo destruction, 2) curettage, 3) photodynamic therapy, 4) surgical excision, 5) topical 5-fluorouracil, 6) topical corticosteroids 7) topical diclofenac, 8) topical imiquimod, 9) topical retinoids, or 10) other treatments for AK including glycolic acid or over-the-counter products containing retinol, alpha or beta hydroxy acids
* Use within 1 month before Visit 1 of 1) immunomodulators or immunosuppressive therapies, 2) interferon, 3) oral or injectable corticosteroids, or 4) cytotoxic drugs
* Known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency
* Inability to understand the requirements of the study and the relative information or are unable or not willing to comply with the study protocol
* Employees of the Investigator or research center or their immediate family members
* Patients who have participated in this study previously
* Patient lived in the same household as currently enrolled subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic equivalence with Reference product | 6 weeks
  Therapeutic equivalence will be evaluated for the primary endpoint at Visit 4 in the PP population. If the 90% confidence interval on the absolute difference between the proportion of subjects who are considered a complete cure in the Test and the Reference product groups (pT - pR) is contained within [-20%, +20%], then therapeutic equivalence of the Test product to the Reference product will be considered to have been demonstrated
Superiority to Placebo | 6 weeks
  The superiority of the Test and Reference products against the Placebo product will be evaluated for the primary endpoint at Visit 4 in the modified Intent-to-Treat (mITT) population using the last observation carried forward (LOCF). If the proportion of subjects who are considered a complete cure in the Test and the Reference product groups is numerically and statistically superior to that of the Placebo (p < 0.05; using a two-sided Cochran-Mantel-Haenszel [CMH] test, stratified by clinical site), then the superiority of the Test and Reference products over Placebo will be concluded
Primary Efficacy End Point | 6 weeks
  The primary efficacy endpoint is the proportion of subjects in each treatment group with treatment success, defined as 100% clearance of all AK lesions (baseline or target AK lesions and any new AK lesions) within the designated treatment area (i.e., complete cure), assessed at study Week 6 (Day 43 ± 4, which is 4 weeks after completion of 2 weeks of treatment)

SECONDARY OUTCOMES:
Safety Analysis | 6 weeks
  All Safety analysis will be based on the Safety population. Adverse events will be classified using standard MedDRA terminology Version 24.0 or higher and summarized by treatment group. Summary tables comparing the type, incidence, date of onset, date of resolution, severity, action taken, outcome, and Investigator's opinion of relationship to the study product will be prepared by treatment group. If sufficient data exist, AE frequencies will be compared between treatments using Fisher's exact test. If the global Fisher's exact test is statistically significant among the three treatment groups at the 5% alpha level (i.e., p < 0.05), then Fisher's exact test using only the Test and Reference groups may be performed to identify any potential statistically significant differences that are clinically relevant between the two active treatment groups

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - CBCC Global Research Site 005, Bakersfield, California
  - CBCC Global Research Site 006, Cerritos, California
  - CBCC Global Research Site 004, Lauderdale Lakes, Florida
  - CBCC Global Research Site 001, Miami, Florida
  - CBCC Global Research Site 002, Miami, Florida
  - CBCC Global Research Site 003, Miramar, Florida
  - CBCC Global Research Site 007, Sugarloaf, Pennsylvania